CLINICAL TRIAL: NCT04214262
Title: A Randomized Phase III Trial of Induction/Consolidation Atezolizumab (NSC #783608) + SBRT Versus SBRT Alone in High Risk, Early Stage NSCLC
Brief Title: Testing the Addition of the Drug Atezolizumab to the Usual Radiation Treatment for Patients With Early Non-small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2019-08627; NCI-2019-08627 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S1914 (Other: SWOG); S1914 (Other: CTEP); U10CA180888 (NIH)
Record Dates: First submitted 2019-12-30; First posted 2020-01-02 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-11

CONDITIONS: Lung Non-Small Cell Carcinoma; Stage I Lung Cancer AJCC v8; Stage II Lung Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — atezolizumab; Specimen Handling; Fluorodeoxyglucose F18; Magnetic Resonance Spectroscopy; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (atezolizumab, SBRT) (Experimental): Patients receive atezolizumab IV over 30-60 minutes on day 1 of each cycle. Treatment repeats every 21 days for 8 cycles in the absence of disease progression or unacceptable toxicity. Starting on day 1 cycle 3, patients also undergo SBRT for 3-8 treatments every 2 days or QD over 1-3 weeks. Patients undergo FDG-PET/CT during screening. Patients undergo blood sample collection and CT scans throughout the trial.
  Interventions: Drug: Atezolizumab; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Other: Fludeoxyglucose F-18; Procedure: Positron Emission Tomography; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Radiation: Stereotactic Body Radiation Therapy
- Arm B (SBRT) (Active Comparator): Beginning 21 days after randomization, patients undergo SBRT for 3-8 treatments every 2 days or QD over 1-3 weeks. Patients undergo FDG-PET/CT during screening. Patients undergo blood sample collection and CT scans throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Other: Fludeoxyglucose F-18; Procedure: Positron Emission Tomography; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Drug: Atezolizumab — Given IV
  Other Names: MPDL 3280A; MPDL 328OA; MPDL-3280A; MPDL3280A; MPDL328OA; RG 7446; RG-7446; RG7446; RO 5541267; RO-5541267; RO5541267; Tecentriq
  Arms: Arm A (atezolizumab, SBRT)
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT or PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Other: Fludeoxyglucose F-18 — Undergo FDG PET/CT
  Other Names: 18FDG; FDG; Fludeoxyglucose (18F); fludeoxyglucose F 18; Fludeoxyglucose F18; Fluorine-18 2-Fluoro-2-deoxy-D-Glucose; Fluorodeoxyglucose F18
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Radiation: Stereotactic Body Radiation Therapy — Undergo SBRT
  Other Names: SABR; SBRT; Stereotactic Ablative Body Radiation Therapy

SUMMARY:
This phase III trial studies how well atezolizumab added to the usual radiation therapy works in treating patients with stage I-IIA non-small cell lung cancer. Immunotherapy with monoclonal antibodies, such as atezolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Radiation therapy, such as stereotactic body radiation therapy, uses special equipment to position a patient and deliver radiation to tumors with high precision. This method can kill tumor cells with fewer doses over a shorter period and cause less damage to normal tissue. Giving atezolizumab and radiation therapy may work better than radiation therapy alone in treating patients with early non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare overall survival (OS) in patients with inoperable, early stage non-small cell lung cancer (NSCLC) randomized to stereotactic body radiation therapy (SBRT) with or without atezolizumab.

SECONDARY OBJECTIVES:

I. To compare investigator-assessed progression-free survival (IA-PFS) between the arms.

II. To compare progression free survival (PFS) by blinded independent centralized review (BIRC) between the arms in a random subset of patients.

III. To evaluate distant, locoregional, and local failure rates within each treatment arm.

IV. To evaluate the frequency and severity of toxicities within each treatment arm.

ADDITIONAL OBJECTIVE:

I. To collect specimens for banking.

HEALTH-RELATED QUALITY OF LIFE (HRQOL) OBJECTIVE:

I. This objective will not be met, as the study was closed following the first interim analysis.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients receive atezolizumab intravenously (IV) over 30-60 minutes on day 1 of each cycle. Treatment repeats every 21 days for 8 cycles in the absence of disease progression or unacceptable toxicity. Starting on day 1 cycle 3, patients also undergo SBRT for 3-8 treatments every 2 days or once daily (QD) over 1-3 weeks. Patients undergo fludeoxyglucose F-18 (FDG)-positron emission tomography/computed tomography (PET/CT) during screening. Patients undergo blood sample collection and CT scans throughout the trial.

ARM B: Beginning 21 days after randomization, patients undergo SBRT for 3-8 treatments every 2 days or QD over 1-3 weeks. Patients undergo FDG-PET/CT during screening. Patients undergo blood sample collection and CT scans throughout the trial.

After completion of study treatment, patients are followed for 5 years after randomization.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have histologically or cytologically proven stage I-IIA or limited T3N0M0 non-small cell lung cancer (NSCLC), without radiographic evidence of nodal or distant involvement (N0M0). Patient may have T3 disease with the exclusion of pericardial involvement. Patients with multifocal tumors with no more than two lesions confirmed or suspected to be synchronous early stage NSCLCs are eligible provided at least one lesion is histologically or cytologically proven to be NSCLC and meets one or more high-risk features
* Disease must have one or more of the following high-risk features:

  * Tumor diameter >= 2 cm (inclusive of any non-solid, ground glass component) as assessed by diagnostic CT
  * Tumor standard uptake value (SUV) max >= 6.2 as assessed by FDG PET/CT
  * Moderately differentiated, poorly differentiated, or undifferentiated histology
* Patient must have undergone diagnostic chest CT with or without contrast (IV contrast preferred) within 42 days prior to randomization. PET-CT may be used if the CT portion is of comparable diagnostic quality to a stand-alone CT. All disease must be assessed within 42 days prior to randomization
* Patient must have undergone FDG PET/CT of chest within 90 days prior to randomization
* Patient must not have evidence of hilar or mediastinal nodal involvement. Any patient with radiographically suspicious hilar or mediastinal nodes (including features such as non-calcified nodes with a short axis diameter > 1 cm, abnormal morphology, and/or elevated FDG avidity) must undergo cytologic sampling of suspicious nodes to rule out involvement prior to randomization. Mediastinal nodal sampling for other patients is optional. For cases in which the treating physician/multidisciplinary opinion is used to define nodes as "non-suspicious" (such as long-standing, stable enlarged nodes from other medical causes), the rationale must be clearly documented within the medical record
* Patient must have undergone history and physical examination within 28 days prior to randomization
* Patient must be medically or surgically inoperable as documented by the evaluating thoracic surgeon or multi-disciplinary tumor board consensus OR patient's unwillingness to undergo surgical resection must be clearly documented
* Patient must not have received any prior treatment for the current NSCLC diagnosis
* Patient must not have undergone prior radiation to overlapping regions of the chest that, in the opinion of the treatment physician, will interfere with protocol treatment
* Patient must not have received treatment with systemic immunostimulatory or immunosuppressive agents, including corticosteroids, within 14 days prior to randomization
* Patient must be >= 18 years old
* Patient must have Zubrod performance status of 0-2
* Patient must have adequate liver function defined as aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 3 x institutional upper level of normal (IULN) within 28 days prior to randomization
* Patient must have adequate renal function defined as calculated creatinine clearance >= 30 mL/min using the following formula. The serum creatinine value used in the calculation must have been collected within 28 days prior to randomization
* Patient must have absolute neutrophil count (ANC), platelets, and hemoglobin measured within 28 days prior to randomization. The purpose of these tests is to collect baseline values to compare with on-treatment values
* Patient must have thyroid-stimulating hormone (TSH) measured within 28 days prior to randomization. The purpose of this test is to collect baseline values to compare with on-treatment values
* Patient must not have significant cardiovascular disease (New York Heart Association [NYHA] class II or greater)
* Patient must not have myocardial infarction within 90 days prior to randomization
* Patient must not have unstable arrhythmias or unstable angina
* Patient must not have known left ventricular ejection fraction (LVEF) < 40% within 28 days prior to randomization

  * NOTE: Assessment of LVEF by echocardiogram or multigated acquisition (MUGA) is not an eligibility requirement, but if a standard of care echocardiogram or MUGA was clinically indicated, the LVEF must not be < 40% within 28 days prior to randomization
* Patient must not have had an infection >= grade 3 (Common Terminology Criteria for Adverse Events [CTCAE] version 5.0) within 28 days prior to randomization
* Patient must not have an active autoimmune disease that has required systemic treatment in past two years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed
* Patient must be tested for hepatitis B within 28 days prior to randomization. Patient must not have active (chronic or acute) hepatitis B virus (HBV) infection. Patients may have past or resolved HBV infection

  * Active HBV is defined as having a positive hepatitis B surface antigen (HBsAg) test
  * Past or resolved HBV is defined as having a negative HBsAG test and a positive total hepatitis B core antibody (HBcAb) test
* Patient must be tested for hepatitis C within 28 days prior to randomization. Patient must not have active hepatitis C virus (HCV) infection

  * Active HCV is defined as having a positive HCV antibody test followed by a positive HCV ribonucleic acid (RNA) test
* Patient must have pulmonary function testing to include, at a minimum, forced expiratory volume in 1 second (FEV1) and Diffusing capability of carbon monoxide (DLCO) documented within 90 days prior to randomization
* Patients with known human immunodeficiency virus (HIV) infection must be receiving anti-retroviral therapy and have an undetectable viral load at their most recent viral load test within 6 months prior to randomization
* Patient must not have a history of clinically significant interstitial lung disease or evidence of active pneumonitis on the screening chest CT
* Patients must not have a prior or concurrent malignancy whose natural history or treatment has the potential (in the opinion of the treating physician) to interfere with the safety or efficacy assessment of the investigational regimen
* Patients must not be pregnant due to the potential teratogenic side effects of the protocol treatment. Women of reproductive potential and men must have agreed to use an effective contraception method for the duration of protocol treatment, and for 5 months (150 days) after the last dose of atezolizumab. A woman is considered to be of "reproductive potential" if she has had a menses at any time in the preceding 12 consecutive months. In addition to routine contraceptive methods, "effective contraception" also includes heterosexual celibacy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) defined as a hysterectomy, bilateral oophorectomy or bilateral tubal ligation. However, if at any point a previously celibate patient chooses to become heterosexually active during the time period for use of contraceptive measures outlined in the protocol, he/she is responsible for beginning contraceptive measures. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with atezolizumab, breastfeeding must be discontinued prior to randomization
* Patients of reproductive potential must have a negative serum pregnancy test within 14 days prior to randomization
* Patients must not have known active tuberculosis
* Patients must not have received a live, attenuated vaccine within 28 days prior to randomization

  * NOTE: All coronavirus disease 2019 (COVID-19) vaccines that have received Food and Drug Administration (FDA) approval or FDA emergency use authorization are acceptable
* Patients must not have a known history of allergic reactions attributed to compounds of similar chemical or biologic composition to atezolizumab
* Patients must not have a known history of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric antibodies, fusion proteins, or Chinese hamster ovary cell products or to any component of the atezolizumab formulation
* Patient must agree to have specimens submitted for translational medicine and banking
* Patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines
* As a part of the OPEN registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system
* Patients who can complete quality of life instruments in English, French, or Spanish must agree to complete the questionnaires at the protocol-specified time points

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2020-08-13 (Actual); Primary Completion 2028-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | From date of randomization to date of death due to any cause, assessed up to 3 years
  Will compare overall survival between patients with inoperable, T1, T2, limited T3, N0M0 (early stage) non-small cell lung cancer randomized to stereotactic body radiation therapy with or without atezolizumab. Will be evaluated using the method of Kaplan-Meier. For point estimates at landmark times, the associated 95% confidence interval (CI) will be calculated using Greenwood's formula and based on a log-log transformation applied on the survival function. Hazard ratios for these outcomes will be estimated using a Cox Proportional Hazards regression model and estimated using a stratified Cox regression model.

SECONDARY OUTCOMES:
Progression free survival | From date of randomization to date of first documentation of progression or death due to any cause, assessed up to 5 years
  Will be evaluated using the method of Kaplan-Meier. For point estimates at landmark times, the associated 95% CI will be calculated using Greenwood's formula and based on a log-log transformation applied on the survival function. Hazard ratios for these outcomes will be estimated using a Cox Proportional Hazards regression model and estimated using a stratified Cox regression model.
Incidence of adverse events | Up to 5 years
  This study will utilize the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 for toxicity and serious adverse event reporting.

OTHER OUTCOMES:
Change in health-related quality of life | Up to 5 years
  As measured by the EORTC Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) and EORTC-QLQ-LC13, between arms. The scores at baseline and subsequent time points, as well the changes from baseline at each time point for each treatment group will be analyzed as continuous variables and compared using the two-sample t-test.

CONTACTS AND LOCATIONS:
Overall Officials: Megan E Daly, Principal Investigator — SWOG Cancer Research Network
Locations (391):
- United States (391):
  - Providence Alaska Medical Center, Anchorage, Alaska
  - NEA Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - AIS Cancer Center at San Joaquin Community Hospital, Bakersfield, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Tower Cancer Research Foundation, Beverly Hills, California
  - Kaiser Permanente Dublin, Dublin, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Veterans Affairs Loma Linda Healthcare System, Loma Linda, California
  - Tibor Rubin VA Medical Center, Long Beach, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Memorial Medical Center, Modesto, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Saint Joseph Hospital - Orange, Orange, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Desert Regional Medical Center, Palm Springs, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - The Permanente Medical Group-Roseville Radiation Oncology, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente Cancer Treatment Center, South San Francisco, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Gene Upshaw Memorial Tahoe Forest Cancer Center, Truckee, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Presbyterian Intercommunity Hospital, Whittier, California
  - Rocky Mountain Regional VA Medical Center, Aurora, Colorado
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Memorial Hospital North, Colorado Springs, Colorado
  - Kaiser Permanente-Franklin, Denver, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Cancer Care and Hematology-Fort Collins, Fort Collins, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - UCHealth Greeley Hospital, Greeley, Colorado
  - UCHealth Highlands Ranch Hospital, Highlands Ranch, Colorado
  - Kaiser Permanente-Rock Creek, Lafayette, Colorado
  - Kaiser Permanente-Lone Tree, Lone Tree, Colorado
  - Medical Center of the Rockies, Loveland, Colorado
  - Banner North Colorado Medical Center - Loveland Campus, Loveland, Colorado
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Smilow Cancer Hospital Care Center at Greenwich, Greenwich, Connecticut
  - Smilow Cancer Hospital Care Center - Guilford, Guilford, Connecticut
  - Smilow Cancer Hospital-Hamden Care Center, Hamden, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - Bayhealth Hospital Kent Campus, Dover, Delaware
  - Beebe South Coastal Health Campus, Millville, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - GenesisCare USA - Aventura FP, Aventura, Florida
  - GenesisCare USA - Aventura, Aventura, Florida
  - Jupiter Medical Center, Jupiter, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Memorial Hospital West, Pembroke Pines, Florida
  - GenesisCare USA - Plantation, Plantation, Florida
  - Florida Cancer Specialists - Sarasota, Sarasota, Florida
  - Florida Cancer Specialists - Sarasota Downtown, Sarasota, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Sarasota Memorial Health Care Center at University Parkway, Sarasota, Florida
  - Augusta Oncology Associates PC-D'Antignac, Augusta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Rush-Copley Medical Center, Aurora, Illinois
  - OSF Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Jesse Brown Veterans Affairs Medical Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - UW Health Carbone Cancer Center Rockford, Rockford, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Community Cancer Center South, Indianapolis, Indiana
  - McFarland Clinic - Ames, Ames, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Saint Joseph Hospital East, Lexington, Kentucky
  - LSU Health Baton Rouge-North Clinic, Baton Rouge, Louisiana
  - Our Lady of the Lake Physician Group, Baton Rouge, Louisiana
  - Louisiana Hematology Oncology Associates LLC, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center - Houma, Houma, Louisiana
  - Terrebonne General Medical Center, Houma, Louisiana
  - East Jefferson General Hospital, Metairie, Louisiana
  - UM Saint Joseph Medical Center, Towson, Maryland
  - Beverly Hospital, Beverly, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - Beth Israel Deaconess Medical Center/Winchester Center for Cancer Care, Winchester, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Michigan Healthcare Professionals Clarkston, Clarkston, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Michigan Healthcare Professionals Farmington, Farmington Hills, Michigan
  - Corewell Health Farmington Hills Hospital, Farmington Hills, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Michigan Healthcare Professionals Macomb, Macomb, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Henry Ford Health Providence Novi Hospital, Novi, Michigan
  - Michigan Healthcare Professionals Pontiac, Pontiac, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Henry Ford Health Providence Southfield Hospital, Southfield, Michigan
  - MyMichigan Medical Center Tawas, Tawas City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Corewell Health Beaumont Troy Hospital, Troy, Michigan
  - Michigan Healthcare Professionals Troy, Troy, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Baptist Memorial Hospital and Cancer Center-Golden Triangle, Columbus, Mississippi
  - Baptist Cancer Center-Grenada, Grenada, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Union County, New Albany, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Freeman Health System, Joplin, Missouri
  - Kansas City Veterans Affairs Medical Center, Kansas City, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Nebraska Medicine-Bellevue, Bellevue, Nebraska
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Capital Health Medical Center-Hopewell, Pennington, New Jersey
  - MD Anderson Cancer Center at Cooper-Voorhees, Voorhees Township, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - New York-Presbyterian/Brooklyn Methodist Hospital, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - Mary Imogene Bassett Hospital, Cooperstown, New York
  - The Cancer Institute at Saint Francis Hospital, East Hills, New York
  - Arnot Ogden Medical Center/Falck Cancer Center, Elmira, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - Mount Sinai Chelsea, New York, New York
  - Mount Sinai West, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Manhattan Eye Ear and Throat Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Lenox Hill Hospital, New York, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Good Samaritan University Hospital, West Islip, New York
  - Messino Cancer Centers, Asheville, North Carolina
  - UNC Health Cancer Care Cary, Cary, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Durham VA Medical Center, Durham, North Carolina
  - UNC Health Cancer Care Garner, Garner, North Carolina
  - CaroMont Regional Medical Center, Gastonia, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Novant Health Cancer Institute - Huntersville, Huntersville, North Carolina
  - Novant Health Cancer Institute - Kernersville, Kernersville, North Carolina
  - Novant Health Cancer Institute - Matthews, Matthews, North Carolina
  - CarolinaEast Medical Center, New Bern, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - UNC Health Cancer Care Raleigh, Raleigh, North Carolina
  - UNC Health Cancer Care Wakefield, Raleigh, North Carolina
  - Novant Cancer Institute Radiation Oncology - Supply, Supply, North Carolina
  - Novant Health Cancer Institute Radiation Oncology - Wilmington, Wilmington, North Carolina
  - Novant Health New Hanover Regional Medical Center, Wilmington, North Carolina
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Miami Valley Hospital South, Centerville, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Premier Blood and Cancer Center, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Mount Carmel Grove City Hospital, Grove City, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - IRMC Cancer Center, Indiana, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - UPMC Cancer Center - Monroeville, Monroeville, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Jefferson Torresdale Hospital, Philadelphia, Pennsylvania
  - UPMC-Saint Margaret, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Geisinger Medical Oncology-Selinsgrove, Selinsgrove, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Saint Joseph's/Candler - Bluffton Campus, Bluffton, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Baptist Memorial Hospital and Cancer Center-Collierville, Collierville, Tennessee
  - Ballad Health Cancer Care - Kingsport, Kingsport, Tennessee
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - MD Anderson in The Woodlands, Conroe, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - MD Anderson West Houston, Houston, Texas
  - MD Anderson League City, League City, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - George E Wahlen Department of Veterans Affairs Medical Center, Salt Lake City, Utah
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Augusta Health Center for Cancer and Blood Disorders, Fishersville, Virginia
  - Ballad Health Cancer Care - Norton, Norton, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - Legacy Cancer Institute Medical Oncology and Day Treatment, Vancouver, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - Wheeling Hospital/Schiffler Cancer Center, Wheeling, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Ascension Saint Elizabeth Hospital, Appleton, Wisconsin
  - Northwest Wisconsin Cancer Center, Ashland, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Elmbrook Campus, Brookfield, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Ascension Calumet Hospital, Chilton, Wisconsin
  - HSHS Sacred Heart Hospital, Eau Claire, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Ascension Saint Francis - Reiman Cancer Center, Franklin, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Bellin Memorial Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Mayo Clinic Health System-Franciscan Healthcare, La Crosse, Wisconsin
  - William S Middleton VA Medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Aspirus Medford Hospital, Medford, Wisconsin
  - Ascension Columbia Saint Mary's Hospital Ozaukee, Mequon, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Ascension Columbia Saint Mary's Hospital - Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - ThedaCare Cancer Care - New London, New London, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Ascension Mercy Hospital, Oshkosh, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Ascension All Saints Hospital, Racine, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Aspirus Cancer Care - James Beck Cancer Center, Rhinelander, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sheboygan, Sheboygan, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Ascension Medical Group Southeast Wisconsin - Mayfair Road, Wauwatosa, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

DOCUMENTS (1):
  • Informed Consent Form (2024-02-23): https://cdn.clinicaltrials.gov/large-docs/62/NCT04214262/ICF_000.pdf